CLINICAL TRIAL: NCT01651754
Title: Humoral and Cellular Immune Responses After Influenza Vaccination in Patients With Postcancer Fatigue and in Patients With Chronic Fatigue Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UMCNONCO201009
Record Dates: First submitted 2012-06-21; First posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-06

CONDITIONS: Postcancer Fatigue; Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Seasonal influenza vaccination (Other)
  Interventions: Biological: Seasonal influenza vaccination

INTERVENTIONS:
Biological: Seasonal influenza vaccination — single dose of influenza vaccination

SUMMARY:
Postcancer fatigue (PCF) is a frequently occurring, severe and invalidating problem, impairing quality of life. Patients with chronic fatigue syndrome (CFS) also suffer from severe fatigue symptoms. Although it is possible to effectively treat CFS, the nature of the underlying physiology remains unclear. The presence of an underlying immunological problem has been suggested as an explanation for PCF and CFS. The aim of this study is to compare the humoral and cellular immune responses upon influenza vaccination in PCF patients, CFS patients, non-fatigued cancer survivors, and healthy controls.

PCF (n=20) and CFS patients (n=20) will be vaccinated against influenza. Age and gender matched non-fatigued cancer survivors (n=20) and healthy controls (n=20) will be included for comparison. Antibody responses will be measured at baseline and at day 21 by a hemagglutination inhibition test. T cell responses will be measured at baseline and at day 7 by lymphocyte proliferation, activation, and cytokine secretion.

DETAILED DESCRIPTION:
Background PCF is a frequently occurring, severe, and invalidating problem in cancer survivors, impairing quality of life. The prevalence of PCF observed in longitudinal follow-up studies ranged from 19-39%. Cognitive behavior therapy, especially designed for PCF, seemed to be an effective treatment option for PCF. However, although it is now possible to effectively treat PCF, the nature of the underlying physiology of PCF remains unclear.

Hypotheses about mechanisms explaining cancer-related fatigue have already been described, including dysregulation of brain serotonin, dysregulation of the hypothalamic-pituitary-adrenal axis responsiveness, disruption of the circadian rhythm, alterations in muscle and ATP metabolism, and activation of the vagal afferent nerve. Furthermore, the presence of an underlying immunological problem has been suggested as an explanation for PCF.

Another group of patients suffering from severe fatigue symptoms are patients with CFS. The estimated worldwide prevalence of CFS is 0.4-1%. In the Netherlands, about 100.000 patients are suffering from chronic fatigue, of which 30.000 to 40.000 suffer from CFS. In contrast to fatigue in patients with PCF, in patients with CFS no clear precipitating factor could be identified. Also for patients with CFS, a cognitive behavior therapy is designed, which is proven to be effective, but the pathophysiological mechanism of CFS remains unclear.

Hypotheses explaining the pathophysiological mechanism of CFS include morphological and metabolic alterations in the brain, diminished central activation of muscles, altered central nervous system functioning, a neuroendocrine disturbance, or cognitive impairment. Furthermore, the presence of an underlying immunological problem has been suggested as an explanation for CFS.

If an underlying immunological problem is present, PCF and CFS patients might have an altered response to vaccination.

Aim Therefore, the aim of this study is to compare the humoral and cellular immune responses upon vaccination, using seasonal influenza vaccination as a model of a vaccination, in PCF and CFS patients, non-fatigued cancer survivors, and healthy controls.

Research questions

1. Is the humoral and/or cellular immune response after influenza vaccination different between fatigued patients (PCF and CFS) and non-fatigued individuals?
2. Is the humoral and/or cellular immune response after influenza vaccination different between PCF and CFS patients? Design The immune responses upon influenza vaccination will be assessed in 20 PCF patients and in 20 CFS patients. As a control group for PCF patients, 20 non-fatigued cancer survivors will be included. Additionally, 20 healthy controls will participate in this study as a control group without a cancer history and without fatigue symptoms. These four groups will be age- and sex-matched.

At baseline, participants will complete the Checklist Individual Strength, a questionnaire about the current use of medicines, and a questionnaire about their vaccination history. All participants will be intramuscularly vaccinated with a single dose of the seasonal influenza vaccine. Peripheral blood mononuclear cells will be collected at baseline (day 1) and 7 days after vaccination (day 8), and serum will be collected at baseline and 21 days after vaccination (day 22). Half a year after vaccination, all participants will be contacted to check whether a possible infection by influenza had taken place in the meantime or not.

The humoral immune responses on influenza vaccination will measured at day 1 and day 22 in serum by the haemagglutination-inhibition antibody test. The cellular immune responses will be measured at day 1 and day 8 by T lymphocyte proliferation, activation, and cytokine secretion.

Relevance of this study To the best of our knowledge, we are the first to explore both the humoral and cellular immune responses after influenza vaccination in both PCF and CFS patients. By means of this study, we would like to improve the understanding of the underlying physiology of PCF and CFS.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria
* Age between 18 and 60 years old
* Written informed consent Inclusion criteria cancer survivors
* Severely fatigued (CIS-fatigue score ≥ 35) or non-fatigued (CIS-fatigue < 27)
* Treated for a malignant, solid tumor
* Completion of treatment for cancer minimal 1 year ago
* Disease-free, as defined by the absence of somatic disease activity parameters
* Age at disease onset minimal 18 years Inclusion criteria CFS patients
* Severe, persistent or continuously returning complaints of fatigue, which do not improve noteworthy after rest and which are not the consequence of continuous exertion
* The fatigue resulted into a substantial decrease in former levels of professional, social and/or personal functioning
* The complaints cannot be explained by a physical cause
* The complaints persist for at least 6 months

Exclusion Criteria:

* - Psychological or psychiatric treatment
* Physical comorbidity that could explain the fatigue
* Treatment with anti-depressive drugs, anti-epileptic drugs, or benzodiazepines
* A known immune deficiency
* Treatment with corticosteroids during the last 2 weeks
* Symptoms of influenza
* Allergy for chicken protein

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Humoral and cellular immune responses after influenza vaccination in patients with postcancer fatigue and in patients with chronic fatigue syndrome. | before vaccination, 1 and 3 weeks after vaccination (change in immune response from pre- to post-vaccination)
  Humoral and cellular immune responses after influenza vaccination in patients with postcancer fatigue and in patients with chronic fatigue syndrome. The humoral immune responses will be measured by the hemagglutination-inhibition antibody test. The cellular immune responses will be measured by T lymphocyte proliferation and cytokine secretion of peripheral blood mononuclear cells. A full blood cell count will be performed and hemoglobin, glucose, and cholesterol levels, iron status, electrolyte balance, erythrocyte sedimentation rate, and thyroid, kidney, and liver function will be checked.

CONTACTS AND LOCATIONS:
Overall Officials: H.W.M. van Laarhoven, Md, Principal Investigator — University Medical Centre Nijmegen st Radboud
Locations (1):
- University Medical Centre Nijmegen st Radboud, Nijmegen, Netherlands